CLINICAL TRIAL: NCT04117386
Title: Prevalence of HPV-associated Eye Infection and Cytokine Levels in Tears From Patients Diagnosed With Pterygium
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Ngamjit Kasetsuwan, Associate professor, Chulalongkorn University
Other Study IDs: IRB NO. 405/62
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Human Papilloma Virus Infection; Pterygium
Keywords: HPV infection; Pterygium; Cytokine; VEGF; auto-inoculation
MeSH Terms: conditions — Papillomavirus Infections; Pterygium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary pterygium group: Participants who was diagnosed with primary pterygium
  Interventions: Diagnostic Test: HPV genotyping assay using HPV GenoArray Diagnostic Kits (Hybribio Ltd., Sheung Wan, Hong Kong); Diagnostic Test: Bio-Plex® 200 system (Bio- Rad, Hercules, CA)
- Secondary pterygium group: Participants who was diagnosed with secondary pterygium
  Interventions: Diagnostic Test: HPV genotyping assay using HPV GenoArray Diagnostic Kits (Hybribio Ltd., Sheung Wan, Hong Kong); Diagnostic Test: Bio-Plex® 200 system (Bio- Rad, Hercules, CA)
- Healthy participants as control group: Participants who have no pterygium and other inflammation disease in eyes
  Interventions: Diagnostic Test: HPV genotyping assay using HPV GenoArray Diagnostic Kits (Hybribio Ltd., Sheung Wan, Hong Kong); Diagnostic Test: Bio-Plex® 200 system (Bio- Rad, Hercules, CA)

INTERVENTIONS:
Diagnostic Test: HPV genotyping assay using HPV GenoArray Diagnostic Kits (Hybribio Ltd., Sheung Wan, Hong Kong) — HPV genotyping assay using HPV GenoArray Diagnostic Kits (Hybribio Ltd., Sheung Wan, Hong Kong) for swab sample collected from pterygium and normal conjunctiva and also for urine collected in Colli-PeeTM device (Novosanis, Belgium)
Diagnostic Test: Bio-Plex® 200 system (Bio- Rad, Hercules, CA) — Bioplex was use for measure cytokine IL-6, IL-18 and VEGF from tears collected from Schirmer strip

SUMMARY:
Prevalence of HPV-associated eye infection and cytokine levels in tears from patients diagnosed with pterygium

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the prevalence of HPV infection in primary and recurrent pterygium and the association of HPV types collecting from conjunctiva swab and urine. The second purpose is to compare a quantity of cytokines including IL-6, IL-18 and growth factor including VEGF found in tears of patients with primary and recurrent pterygium to participants with free of ocular disease Primary hypothesis

- The prevalence of HPV infection in primary pterygium is difference with prevalence in recurrent pterygium patients.

Secondary hypothesis

* Ocular HPV infection has association with HPV genitalia infection.
* Tears cytokine and growth factor level (IL-6, IL-18 and VEGF) are higher in pterygium HPV infection than non-HPV infection and also more than normal population

ELIGIBILITY:
Participants as primary and secondary pterygium group

Inclusion Criteria:

* Age above 18 years old
* presence of pterygium invading the cornea

Exclusion Criteria:

* Other ocular inflammation that could affect the results of the study (such as conjunctivitis, keratitis, conjunctival tumor, etc) or would preclude the enrollment for safety reasons

Participant without ocular disease Inclusion criteria

* Age above 18 years old Exclusion criteria
* Presence of any ocular inflammation diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population:Patients diagnosed with primary pterygium and recurrent pterygium Target Population: Patients diagnosed with primary pterygium at out-patient clinic, Department of Ophthalmology, King Chulalongkorn Memorial Hospital Control Population: participants without any ocular diseases
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
HPV prevalence | 1 hour per participants which is on a day for collecting sample
  1. To compare HPV prevalence in subjects with primary pterygium and with recurrent pterygium

SECONDARY OUTCOMES:
HPV autoinoculation | 1 hour per participants which is on a day for collecting sample
  To assess whether HPV autoinoculation is present, we evaluate whether there is an association between HPV ocular infection and genital infection.
cytokine IL-6, IL-18 and VEGF levels | 1 hour per participants which is on a day for collecting sample
  To compare cytokine IL-6, IL-18 and VEGF levels among various subgroups, including recurrent pterygium subjects with HPV positive and HPV negative status, primary pterygium subjects with HPV positive and HPV negative, and subjects without ocular diseases

CONTACTS AND LOCATIONS:
Overall Officials: Ngamjit Kasetsuwan, Principal Investigator — Department of Ophthalmology, Chulalongkorn University
Locations (1):
- Faculty of medicine, Chulalongkorn university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
If there is anybody contacting our team for data in the purpose of future research, we agree to share our data.
Supporting Information: Study Protocol, CSR
Time Frame: 1 year after published